CLINICAL TRIAL: NCT01121835
Title: A 24-week, Open, Multicenter, Comparative Study of 2 Strategies (Including Insulin Glargine Versus Premixed Insulin) for the Therapeutic Management of Patients With Type 2 Diabetes Failing Oral Agents
Brief Title: Insulins Glargine and gluLisine strAtegy Versus Premixed Insulin strAteGy: a cOmparative Study
Acronym: GALAPAGOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_C_04589; 2009-018172-33 (EudraCT Number); U1111-1116-9859 (Other: UTN)
Record Dates: First submitted 2010-05-06; First posted 2010-05-12 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine

ARMS (2):
- Insulin glargine (Experimental): Administered once a day in the evening, at the same time every day. The starting daily dose is 0.2 U/Kg of body weight or 12 U, at the investigator's decision.
  Insulin glulisine is administered for patients of the insulin glargine group requiring insulin glulisine at week 12 (visit 11).
  Insulin glulisine is administered prior (10-15 min) to the main meal of the day, which is the meal with highest Post-Prandial Plasma Glucose (PPPG) on the 3 profiles performed before week 12.
  Starting dose is of 4 units per day.
  Interventions: Drug: INSULIN GLARGINE; Drug: INSULIN GLULISINE
- Premixed insulin (Experimental): administered once a day (in the evening at dinner) or twice a day (in the morning before breakfast and in the evening at dinner). Starting daily dose will be 6 U at breakfast and 6 U at dinner, if administered twice a day or 12 U at dinner if administered once a day
  Interventions: Drug: PREMIXED INSULIN

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: solution for injection Route of administration: sub-cutaneous injection Dose regimen: 100 Units/mL solution for injection in a pre-filled SoloStar pen (3 ml)
  Arms: Insulin glargine
Drug: INSULIN GLULISINE — Pharmaceutical form: solution for injection Route of administration: sub-cutaneous Dose regimen: 100 Units/mL solution for injection in a pre-filled SoloStar pen (3 mL)
  Arms: Insulin glargine
Drug: PREMIXED INSULIN — Pharmaceutical form: solution for injection Route of administration: sub-cutaneous Dose regimen: - 30% soluble insulin aspart and 70 % protamine-crystallised insulin aspart in pre-filled Flexpen for all the countries except Mexico
  * 25 % insulin lispro solution and 75% insulin lispro protamine in cartridges for Humapen Luxura for Mexico only
  Arms: Premixed insulin

SUMMARY:
Primary Objective:

To demonstrate the superiority of a strategy with insulin glargine in comparison with a strategy including the premixed insulin in term of percentage of patients reaching HbA1c (glycosylated hemoglobin) below 7% at the end of treatment and who do not experience documented symptomatic hypoglycemia (confirmed by a Plasma Glucose (PG) below 56 mg/dL (3.1 mmol/L)) over a 24-week treatment period, in Type 2 diabetes patients failing lifestyle management and oral agents.

Secondary Objectives:

To assess the effect of insulin glargine in comparison with premixed insulin on :

* Evolution of HbA1c level during the treatment period Percentage of patients who reach the target of HbA1c < 7 % and who do not experience documented symptomatic hypoglycemia confirmed by a Plasma Glucose (PG) below 70 mg/dL (3.9 mmol/L)
* Percentage of patients who reach the target of HbA1c < 6.5% and who do not experience documented symptomatic hypoglycemia confirmed by a PG below 56 mg/dL (3.1 mmol/L) >Percentage of patients who reach the target of HbA1c < 6.5% and who do not experience documented symptomatic hypoglycemia confirmed by a PG below 70 mg/dL (3.9 mmol/L) >Evolution of Fasting Plasma Glucose Evolution of 7-point plasma glucose profiles
* Evolution of weight
* Hypoglycemia occurrence
* Dose of insulins
* Evolution of liver function
* Overall safety

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes diagnosed for more than 1 year
* Insulin naïve
* Treated with lifestyle interventions and oral antidiabetic drugs, at least metformin at the maximum tolerated dose (with a minimum dose of 1g/day), for at least 3 months
* HbA1c ≥ 7.0 % and ≤ 10.5%
* Body mass index (BMI) ≤ 40 kg/m2
* Ability and willingness to perform plasma glucose (PG) monitoring using the sponsor-provided glucose meter and to complete the patient diary
* Willingness and ability to comply with the study protocol
* Signed informed consent obtained prior any study procedure

Exclusion criteria:

* Treatment with glucagon-like peptide-1 (GLP-1) agonists in the 3 months prior to study entry
* Previous treatment with insulin (except for treatment of gestational diabetes or brief treatment with insulin for less than 1 week)
* Diabetes other than type 2 diabetes (e.g. type 1 diabetes, diabetes secondary to pancreatic disorders, drug or chemical agent intake)
* Pregnant or lactating women (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method)
* Hospitalized patient (except for routine diabetes check-up)
* Active proliferative retinopathy, as defined by a photocoagulation or vitrectomy occurrence in the 6 months prior to study entry, or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgical treatment during the study, documented by retina examination, in the 2 years prior to study entry
* History of sensitivity to the study drugs or to drugs with a similar chemical structure
* Impaired renal function: creatinine clearance < 60ml/min
* Impaired liver function (ALT, AST > 3 x upper limit of normal range)
* Severe gastro-intestinal disease
* Treatment with corticosteroids with potential systemic action within the 3 months prior to study entry
* Likelihood of requiring treatments during the study which are not permitted
* Treatment with an investigational product in the 30 days prior to study entry
* Alcohol or drug abuse within the last 5 years

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 934 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Glycosylated Haemoglobin (HbA1c) <7% with no documented symptomatic hypoglycemia (confirmed by a Plasma Glucose (PG) ≤ 56 mg/dL [3.1 mmol/L] | From baseline (visit 2, week 0) to visit 14 (week 24)

SECONDARY OUTCOMES:
7-point plasma glucose (PG) profile recorded on 3 consecutive days | From baseline (visit 2, week 0) to visit 14 (week 24)
Self-monitored PG (Plasma Glucose) values over 3 consecutive days | before visit 4 (week 2)
Self-monitored PG (Plasma Glucose) values over 3 consecutive days | before visit 8 (week 6)
Self-monitored PG (Plasma Glucose) values over 3 consecutive days | before visit 12 (week 16)
Weight and supine blood pressure | From baseline (visit 2, week 0) to visit 14 (week 24)
Insulin doses of the day before each visit | from visit 3 (week 1) to visit 14 (week 24)
Biochemistry and lipid profile | From baseline (visit 2, week 0) to visit 14 (week 24)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (96):
- Austria (4):
  - Investigational Site Number 040-004, Sankt Stefan
  - Investigational Site Number 040-002, Vienna
  - Investigational Site Number 040-001, Vienna
  - Investigational Site Number 040-003, Vienna
- Brazil (5):
  - Investigational Site Number 076002, Belém
  - Investigational Site Number 076005, Curitiba
  - Investigational Site Number 076004, Fortaleza
  - Investigational Site Number 076001, Porto Alegre
  - Investigational Site Number 076003, São Paulo
- China (12):
  - Investigational Site Number 156004, Beijing
  - Investigational Site Number 156005, Beijing
  - Investigational Site Number 156006, Beijing
  - Investigational Site Number 156011, Chongqing
  - Investigational Site Number 156009, Dalian
  - Investigational Site Number 156008, Guangzhou
  - Investigational Site Number 156012, Haikou
  - Investigational Site Number 156007, Nanjing
  - Investigational Site Number 156001, Shanghai
  - Investigational Site Number 156002, Shanghai
  - Investigational Site Number 156003, Shanghai
  - Investigational Site Number 156010, Shenyang
- Colombia (5):
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170002, Bogotá
  - Investigational Site Number 170003, Bucaramanga
  - Investigational Site Number 170005, Manizales
  - Investigational Site Number 170004, Pereira
- Denmark (3):
  - Investigational Site Number 208-001, Hvidovre
  - Investigational Site Number 208-003, København NV
  - Investigational Site Number 208-002, København S
- Greece (10):
  - Investigational Site Number 300006, Alexandroupoli
  - Investigational Site Number 300001, Athens
  - Investigational Site Number 300002, Athens
  - Investigational Site Number 300003, Athens
  - Investigational Site Number 300004, Athens
  - Investigational Site Number 300005, Irakleio
  - Investigational Site Number 300011, Maroussi, Athens
  - Investigational Site Number 300008, Thessaloniki
  - Investigational Site Number 300010, Thessaloniki
  - Investigational Site Number 300007, Thessaloniki
- India (7):
  - Investigational Site Number 356008, Bangalore
  - Investigational Site Number 356003, Bangalore
  - Investigational Site Number 356007, Bangalore
  - Investigational Site Number 356006, Bhubaneshwar
  - Investigational Site Number 356001, Hyderabad
  - Investigational Site Number 356005, Hyderabad
  - Investigational Site Number 356004, Trivandrum
- Italy (10):
  - Investigational Site Number 380-010, Catania
  - Investigational Site Number 380-008, Catania
  - Investigational Site Number 380-006, Colleferro
  - Investigational Site Number 380-007, Foggia
  - Investigational Site Number 380-005, Forlì
  - Investigational Site Number 380-001, Genova
  - Investigational Site Number 380-011, Merano
  - Investigational Site Number 380-009, Napoli
  - Investigational Site Number 380-012, Napoli
  - Investigational Site Number 380-004, Parma
- Investigational Site Number 001, Kuwait City, Kuwait
- Mexico (5):
  - Investigational Site Number 484004, Aguascalientes
  - Investigational Site Number 484001, Aguascalientes
  - Investigational Site Number 484003, Guadalajara
  - Investigational Site Number 484002, Guadalajara
  - Investigational Site Number 484005, Puebla City
- Romania (3):
  - Investigational Site Number 642001, Iași
  - Investigational Site Number 642002, Iași
  - Investigational Site Number 642003, Oradea
- South Korea (4):
  - Investigational Site Number 410004, Ansan-si, Kyouggi-do
  - Investigational Site Number 410003, Koyang-si
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410002, Seoul
- Spain (9):
  - Investigational Site Number 724001, Ávila
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724008, Galdakao
  - Investigational Site Number 724007, Lugo
  - Investigational Site Number 724004, Madrid
  - Investigational Site Number 724009, Pamplona
  - Investigational Site Number 724005, Santa Coloma de Gramanet
  - Investigational Site Number 724003, Seville
  - Investigational Site Number 724006, Valencia
- Taiwan (8):
  - Investigational Site Number 158004, Changhua County
  - Investigational Site Number 158007, Kaohsiung Hsien,
  - Investigational Site Number 158006, New Taipei City
  - Investigational Site Number 158001, Taichung
  - Investigational Site Number 158009, Taichung
  - Investigational Site Number 158005, Tainan
  - Investigational Site Number 158002, Taipei
  - Investigational Site Number 158003, Xindian District
- Turkey (Türkiye) (9):
  - Investigational Site Number 792-013, Ankara
  - Investigational Site Number 792-009, Çanakkale
  - Investigational Site Number 792-006, Diyarbakır
  - Investigational Site Number 792-004, Istanbul
  - Investigational Site Number 792-001, Izmir
  - Investigational Site Number 792-016, Konya
  - Investigational Site Number 792-007, Sivas
  - Investigational Site Number 792-005, Trabzon
  - Investigational Site Number 792-002, Van
- Investigational Site Number 784-001, Dubai, United Arab Emirates